CLINICAL TRIAL: NCT04994925
Title: The Effects of Ready Meal Consumption on Self-reported Appetite Ratings and Subsequent Food Intake in Females
Brief Title: Ready Meal Consumption, Appetite and Food Intake in Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Dr. Sangeetha Thondre, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0119_44
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control ready meal (Active Comparator): Control supermarket brand ready meal with high energy density
  Interventions: Other: Control ready meal
- Test ready meal with low energy density (Experimental): Slimming world test ready meal with low energy density
  Interventions: Other: Test ready meal

INTERVENTIONS:
Other: Control ready meal — Supermarket brand lasagne ready meal
  Arms: Control ready meal
Other: Test ready meal — The Slimming World lasagne ready meal
  Arms: Test ready meal with low energy density

SUMMARY:
Overweight and obesity are public health concerns and there is a forecast rise in the consumption of ready meals that are generally high in saturated fat and low in fibre. Slimming World, a commercial weight management organisation has designed a range of ready meals in line with their weight management programme, which advocates an unrestricted intake of low energy dense food in order to aid in weight loss. Hence, it is valuable to understand the satiating properties of ready meals in order to establish if specific ready meals can enhance satiety and contribute to reducing subsequent energy intake. This study aims to explore the effect of ready meals on short-term satiety and food intake among females with a BMI ≥ 25 kg/m2.

DETAILED DESCRIPTION:
A total of 26 female participants aged between 18-65 years attended Oxford Brookes Centre for Nutrition and Health for two separate testing days. The study aimed to investigate the effects of energy matched ready meals (calorie-matched but differing quantities of protein and fat) on appetite and subsequent energy and macronutrient intake. The ready meals (Control = supermarket brand and Test = Slimming World) differed in energy density and macronutrient composition, with satiety responses investigated in the studies. The participants consumed a standard breakfast and four hours later consumed either a test ready meal (lasagne, higher energy density) or the control ready meal (lower energy density). Four hours after lunch participants food intake was measured during an ad libitum buffet tea. Additionally, satiety measurements were recorded using visual analogue scales throughout and participants completed a weighed food diary for the remainder of the test day.

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-smoking females aged between 18-65 years with a BMI ≥ 25 kg/m2.

  * had no known food allergies to the study foods,
  * had no eating disorders,
  * were not following a special diet (e.g. vegetarian, halal),
  * were not taking any medication or supplements known to affect appetite or weight within the month prior to and/or during the study,
  * were not pregnant, planning to become pregnant or breastfeeding,
  * had not significantly changed their physical activity in the 2-4 weeks prior to the study or who did not intend on changing them during the study,
  * were not receiving systemic or local treatment likely to interfere with the evaluation of the study parameters,

Exclusion Criteria:

* females aged below 18 and above 65 years
* BMI less than 25 kg/m2.
* smokers

  * had food allergies to the study foods,
  * had eating disorders,
  * were following a special diet (e.g. vegetarian, halal),
  * were taking any medication or supplements known to affect appetite or weight within the month prior to and/or during the study,
  * were pregnant, planning to become pregnant or breastfeeding,
  * had significantly changed their physical activity in the 2-4 weeks prior to the study or who did not intend on changing them during the study,
  * were receiving systemic or local treatment likely to interfere with the evaluation of the study parameters,
  * had a gastric band/had undergone gastric bypass treatment
  * and/or females who worked in appetite or feeding related areas.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale measurements for Hunger | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means worse outcome.
Visual Analogue Scale measurements for Fullness | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means better outcome.
Visual Analogue Scale measurements for Desire to Eat | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means worse outcome.
Visual Analogue Scale measurements for Prospective Food Consumption | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means worse outcome.
Energy intake after ad libitum buffet tea | 4 hours
  Total energy consumed at the ad libitum tea given 4 hours after the control/test ready meal
Macronutrient intake after ad libitum buffet tea | 4 hours
  Total macronutrient amounts consumed at the ad libitum tea given 4 hours after the control/test ready meal

SECONDARY OUTCOMES:
Visual Analogue Scale measurements of thirst | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means worse outcome.
Visual Analogue Scale measurements of nausea | 9 hours
  Ratings were established prior to breakfast (fasted), then every 30 minutes from commencing breakfast (8 am) until lunch (12 pm). Visual Analogue Scale ratings continued every 15 minutes from commencing lunch until the buffet tea (4 pm), with the last rating being made after finishing the buffet tea. Minimum value 0 mm; maximum value 100 mm; A higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hillier, PhD, Study Director — Solent University
Locations (1):
- Oxford Brookes Centre for Nutrition and Health, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data is confidential and owned by the Study Sponsor and Collaborator.